CLINICAL TRIAL: NCT02007356
Title: A Phase I/II Single-center Study to Assess Safety and Feasibility of Direct Infusions of Donor-derived Virus-specific T-cells in Recipients of Hematopoietic Stem Cell Transplantation With Post-transplant Viral Infections Using the Cytokine Capture System®
Brief Title: A Study to Assess Safety and Feasibility of Direct Infusions of Donor-derived Virus-specific T-cells in Recipients of Hematopoietic Stem Cell Transplantation With Post-transplant Viral Infections Using the Cytokine Capture System®
Acronym: CCS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EKBB 205/13; me12Khanna
Record Dates: First submitted 2013-11-26; First posted 2013-12-10 (Estimated); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Adenovirus Infection; EBV; Cytomegalovirus Infections; Cytokine Capture System; Allogenic Disease
MeSH Terms: conditions — Adenoviridae Infections; Cytomegalovirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- allogeneic HSCT (Experimental): The present study will evaluate and validate in a single-center, open-label, single arm fashion the safety and feasibility of direct infusions of donor-derived pathogen-specific IFN-γ positive T-cells in recipients of HSCT with post-transplant viral infection according to the previously clinically certified CCS® [3-6]. The Investigator will first generate and apply IFN-γ positive selected T-cells to recipients of HSCT with CMV, EBV or adenovirus as previously published. The Investigator aim is to include 6 patients from the University Hospital of Basel.
  With confirmed safety the investigator will in the future perform an efficacy study and extend this treat-ment for other clinically relevant pathogens including human herpesvirus (HHV)-6, HHV-8, polyomaviruses JC and BK and fungi including Aspergillus fumigatus and Candida albicans, to other immunosuppressed patients such as solid organ transplant (SOT) recipients.
  Interventions: Biological: IFN-γ positive selected T-cells

INTERVENTIONS:
Biological: IFN-γ positive selected T-cells

SUMMARY:
To assess the feasibility of donor-derived interferon (IFN)-γ positive select-ed virus-specific T-cells using the cytokine capture system® (CCS) and the safety of subsequent infusion in recipients of hematopoietic stem cell transplantation (HSCT) with treatment refractory post-transplant viral infections. The CCS has already been successfully used in clinical studies in Germany and United Kingdom (UK).

ELIGIBILITY:
Inclusion Criteria:

* Adults > 18 years of age
* Undergone allogeneic HSCT
* Written informed consent
* Patients with treatment refractory infections with adenovirus, cytomegalovirus (CMV) or Epstein-Barr virus (EBV) will be included in case of fulfilling following criteria:

Patient with Adenovirus Infection:

1. Antiviral treatment with cidofovir for at least 7 days

   * no virus load decrease ( ≤ 1 log) or virus load increase on treatment for at least 7 days or
   * cluster of differentiation 3 (CD3) + cells < 300/µL on treatment for at least 7 days
2. Or if antiviral treatment is contraindicated

Patient with EBV:

1. After receipt of at least one anti-cluster of differentiation 20 antigen (CD20)-antibody treat-ment (375 mg/m2)

* No Virus load decrease (≤ 1 log) or virus load increase 7 days after receipt of treatment or
* CD3+ cells < 300/µL 7 days after receipt of treatment or
* Clinical progression

Patient with CMV:

1. Antiviral treatment with ganciclovir or foscavir for 14 days

   - No Virus load decrease (≤ 1 log) or virus load increase on day 14
2. Or if > 2 recurrences despite antiviral treatment with ganciclovir or foscavir for 14 days and CD3+ cells < 300/µL
3. Or if antiviral treatment is contraindicated -

Patient Exclusion Criteria:

* graft-versus-host disease (GVHD) > grade 2 at the time point of planned infusion
* Known allergy to iron-dextran or murine antibodies

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-12 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Level of enriched IFN-γ+ T-cells | 7 days

SECONDARY OUTCOMES:
Treatment efficacy | 7 days
  Treatment efficacy defined as reduction of virus load, in vivo expansion of antigen-specific T cells in peripheral blood as well as reduction of clinical signs of specific viral infection

CONTACTS AND LOCATIONS:
Overall Officials: Nina Khanna, Dr., Principal Investigator — Universitätsspital Basel, Klinik für Infektiologie
Locations (1):
- Universitätsspital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kaufmann GR, Khanna N, Weber R, Perrin L, Furrer H, Cavassini M, Ledergerber B, Vernazza P, Bernasconi E, Rickenbach M, Hirschel B, Battegay M; Swiss HIV Cohort Study. Long-term virological response to multiple sequential regimens of highly active antiretroviral therapy for HIV infection. Antivir Ther. 2004 Apr;9(2):263-74. PMID 15134189